CLINICAL TRIAL: NCT01219699
Title: A Phase IA, Multicenter, Open-label Dose Escalation Study of Oral BYL719, in Adult Patients With Advanced Solid Malignancies, Whose Tumors Have an Alteration of the PIK3CA Gene
Brief Title: A Study of BYL719 in Adult Patients With Advanced Solid Malignancies, Whose Tumors Have an Alteration of the PIK3CA Gene
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBYL719X2101; 2010-018782-32 (EudraCT Number)
Record Dates: First submitted 2010-10-06; First posted 2010-10-13 (Estimated); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Advanced Solid Tumors With an Alteration of the PIK3CA Gene; Estrogen Receptor Positive Breast Cancer
Keywords: advanced solid tumors; mutation; amplification; wild type; PIK3CA gene; dose-escalation; estrogen receptor positive breast cancer
MeSH Terms: interventions — Alpelisib; Fulvestrant

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BYL719 (Experimental): In adult patients with advanced solid malignancies whose tumors have an alteration (mutation or amplification) of the PIK3CA gene, and in patients whose tumors are have wild-type PIK3CA gene
  Interventions: Drug: BYL719
- BYL719 + fulvestrant (Experimental): In post-menopausal patients with estrogen receptor positive locally advanced or metastatic breast cancer whose tumors have an alteration of the PIK3CA gene, and in patients whose tumors are have wild-type PIK3CA gene
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: BYL719 — BYL719 is an oral α-specific phosphatidylinositol-3-kinase (PI3K) inhibitor.
  Arms: BYL719
Drug: Fulvestrant — In adult patients with advanced solid malignancies whose tumors have an alteration (mutation or amplification) of the PIK3CA gene.
  Fulvestrant is an estrogen receptor antagonist, administered by monthly intramuscular injection
  Arms: BYL719 + fulvestrant

SUMMARY:
This is a first-in-man trial, in which BYL719 will be administered to adult patients with advanced solid tumors, whose tumors have an alteration of the PIK3CA gene and whose disease has progressed despite standard therapy or for whom no standard therapy exists. A combination of BYL719 with fulvestrant will also be investigated in post-menopausal patients with locally advanced or metastatic breast cancer whose tumors have an alteration of the PIK3CA gene. The single agent MTD dose expansion cohort and the fulvestrant combination MTD dose expansion cohort will also include ER+/HER2- breast cancer patients whose tumors have the wild type PIK3CA gene

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically-confirmed, advanced unresectable solid tumors who have progressed within three months before screening/baseline visit Only patients who have confirmed PIK3CA status (wild type, mutation or amplification) will be allowed for screening (patients participating in the combination arm must be eligible for treatment with fulvestrant)
* Availability of a representative formalin fixed paraffin embedded tumor tissue sample
* At least one measurable or non-measurable lesion
* Age ≥ 18 years
* World Health Organization (WHO) Performance Status ≤ 2
* Good organ (hepatic, kidney, BM) function at screening/baseline visit

Exclusion Criteria:

* Brain metastasis unless treated and free of signs/symptoms attributable to brain metastasis in the absence of corticosteroid therapy (anti-epileptic therapy is allowed).
* Prior treatment with PI3K, AKT or mTOR inhibitor and failure to benefit
* Patient with peripheral neuropathy NCI-CTC Grade ≥ 3
* Patient with diarrhea NCI-CTC Grade ≥ 2
* Patient with acute or chronic pancreatitis
* Impaired cardiac function or clinically significant cardiac disease incl. unstable angina pectoris ≤ 3 months prior to starting study drug and Acute Myocardial Infarction (AMI) ≤ 3 months prior to starting study drug.
* Patients with clinically manifest diabetes mellitus, history of gestational diabetes mellitus or documented steroid-induced diabetes mellitus
* Women who are pregnant or breast feeding or adults of reproductive potential not employing an effective method of birth control

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2010-10-05 (Actual); Primary Completion 2015-02-05 (Actual); Study Completion 2020-04-16 (Actual)

PRIMARY OUTCOMES:
Incidence rate of dose limiting toxicities (DLT). | 5 years
  MTD (or RP2D) of oral BYL719 as single agent and in combination with fulvestrant.

SECONDARY OUTCOMES:
Overall safety and tolerability of BYL719 as single agent and in combination with fulvestrant | 10 years
  Safety and tolerability: type, intensity, severity and seriousness of adverse events (AE) according to NCI CTCAE v. 4.0.
PK parameters of BYL719 as single agent and in combination with fulvestrant - AUC-tlast and AUC0-inf. | 5 years
  PK parameters AUC-tlast and AUC0-inf
PK parameters of BYL719 as single agent and in combination with fulvestrant - Cmax. | 5 years
  PK parameter Cmax
Pharmacokinetics of BYL719 as single agent and in combination with fulvestrant - Tmax. | 5 years
  PK parameter Tmax
Pharmacokinetics of BYL719 as single agent and in combination with fulvestrant - CL/F. | 5 years
  PK parameter CL/F
Pharmaconkinetics of BYL719 as single agent and in combination with fulvestrant - Vz/F. | 5 years
  PK parameter Vz/F
Pharmacokinetics of BYL719 as single agent and in combination with fulvestrant - Terminal half-life (t1/2) | 5 years
  PK parameter t1/2
Preliminary efficacy of BYL719 as single agent and in combination with fulvestrant by measuring ORR. | 5 years
  Objective tumor response rate (ORR), defined as the sum of complete response and partial response as best reported response by RECIST 1.0 criteria (Novartis v2.0 guideline)
Progression-free survival at maximum tolerated dose | 5 years
  PFS at MTD

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- United States (5):
  - UCSF Medical Center, San Francisco, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Sarah Cannon Research Institute Dept.ofSarahCannonCancerCtr(4), Nashville, Tennessee
  - Vanderbilt Univeristy SC, Nashville, Tennessee
  - MD Anderson Cancer Center/University of Texas MD Anderson, Houston, Texas
- Germany (2):
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Würzburg
- Novartis Investigative Site, Amsterdam, Netherlands
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
- Novartis Investigative Site, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodon J, Demanse D, Rugo HS, Burris HA, Simo R, Farooki A, Wellons MF, Andre F, Hu H, Vuina D, Quadt C, Juric D. A risk analysis of alpelisib-induced hyperglycemia in patients with advanced solid tumors and breast cancer. Breast Cancer Res. 2024 Mar 4;26(1):36. doi: 10.1186/s13058-024-01773-1. PMID 38439079
- [Derived] Juric D, Janku F, Rodon J, Burris HA, Mayer IA, Schuler M, Seggewiss-Bernhardt R, Gil-Martin M, Middleton MR, Baselga J, Bootle D, Demanse D, Blumenstein L, Schumacher K, Huang A, Quadt C, Rugo HS. Alpelisib Plus Fulvestrant in PIK3CA-Altered and PIK3CA-Wild-Type Estrogen Receptor-Positive Advanced Breast Cancer: A Phase 1b Clinical Trial. JAMA Oncol. 2019 Feb 1;5(2):e184475. doi: 10.1001/jamaoncol.2018.4475. Epub 2019 Feb 14. PMID 30543347
- [Derived] Juric D, Rodon J, Tabernero J, Janku F, Burris HA, Schellens JHM, Middleton MR, Berlin J, Schuler M, Gil-Martin M, Rugo HS, Seggewiss-Bernhardt R, Huang A, Bootle D, Demanse D, Blumenstein L, Coughlin C, Quadt C, Baselga J. Phosphatidylinositol 3-Kinase alpha-Selective Inhibition With Alpelisib (BYL719) in PIK3CA-Altered Solid Tumors: Results From the First-in-Human Study. J Clin Oncol. 2018 May 1;36(13):1291-1299. doi: 10.1200/JCO.2017.72.7107. Epub 2018 Feb 5. PMID 29401002
- [Derived] Vora SR, Juric D, Kim N, Mino-Kenudson M, Huynh T, Costa C, Lockerman EL, Pollack SF, Liu M, Li X, Lehar J, Wiesmann M, Wartmann M, Chen Y, Cao ZA, Pinzon-Ortiz M, Kim S, Schlegel R, Huang A, Engelman JA. CDK 4/6 inhibitors sensitize PIK3CA mutant breast cancer to PI3K inhibitors. Cancer Cell. 2014 Jul 14;26(1):136-49. doi: 10.1016/j.ccr.2014.05.020. Epub 2014 Jul 4. PMID 25002028